CLINICAL TRIAL: NCT07384611
Title: Prediction of Difficult Airway in Pediatric Patients Using Preoperative Clinical Parameters
Brief Title: Preoperative Prediction of Difficult Airway in Children
Status: Recruiting | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Sule Ozdemir, Principal İnvestigator, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK-2026-009
Record Dates: First submitted 2026-01-18; First posted 2026-02-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Anesthesia; Difficult Laryngoscopy
Keywords: Pediatric Anesthesia; Difficult Laryngoscopy; Difficult Airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Preoperative Clinical Airway Assessment — Preoperative clinical airway assessment including bedside airway examination and anthropometric measurements performed as part of routine anesthetic evaluation, without any additional intervention beyond standard clinical practice.

SUMMARY:
This prospective observational study aims to evaluate the predictive value of preoperative clinical airway assessment parameters for difficult airway management in pediatric patients undergoing elective surgery under general anesthesia. Preoperative clinical measurements and bedside airway tests will be recorded, and their association with intraoperative airway outcomes, including difficult laryngoscopy and difficult intubation, will be analyzed. Difficult laryngoscopy will be defined as Cormack-Lehane grade III-IV, while secondary outcomes will include difficult intubation, difficult mask ventilation, and airway-related complications. The study seeks to identify clinically applicable predictors and improve preoperative risk stratification for pediatric airway management. The findings may contribute to safer anesthetic practice in children by facilitating early identification of patients at increased airway risk.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 0-12 years
* Scheduled for elective surgery requiring endotracheal intubation under general anesthesia
* ASA physical status I-III
* Written informed consent obtained from parent(s) or legal guardian(s)

Exclusion Criteria:

* Patients older than 12 years
* ASA physical status IV or higher
* Emergency situations that do not allow systematic documentation of the airway management process
* Presence of a congenital or acquired tracheostomy
* Surgical procedures planned to be performed using a supraglottic airway without endotracheal intubation
* Surgical procedures planned to be performed using face mask ventilation without endotracheal intubation
* Inability to obtain parental or legal guardian consent

Ages: 1 Day to 12 Years | Sex: All
Age Groups: Child
Study Population: The study population consists of pediatric patients aged 0 to 12 years who are scheduled for elective surgery under general anesthesia requiring endotracheal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Difficult Laryngoscopy | Perioperative/Periprocedural
  Difficult laryngoscopy defined as Cormack-Lehane grade III or IV during laryngoscopy at tracheal intubation.

SECONDARY OUTCOMES:
First-Attempt Intubation Success | Perioperative/Periprocedural
  Successful tracheal intubation achieved on the first attempt without the need for additional airway devices or techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)